CLINICAL TRIAL: NCT05444491
Title: Based on the Application of Peripheral Blood Polygene Methylation Markers in Postoperative Recurrence Monitoring of Colorectal Cancer
Brief Title: Application of Polygenic Methylation Markers in Postoperative Recurrence Monitoring of Colorectal Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: Singlera Genomics Inc. (Industry)
Collaborators: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: Protector-C
Record Dates: First submitted 2022-06-25; First posted 2022-07-06 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Colorectal Cancer
Keywords: ctDNA methylation; Recurrence monitoring
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MRD positive group: ColonAiQ polygene methylation test was performed on peripheral blood plasma samples from the enrolled patients 4 weeks after surgery. If gene methylation levels in the samples exceeded the threshold, the patients were enrolled in the MRD positive group. The 2-year total tumor recurrence rate of patients in the MRD positive group was calculated, and the positive prediction rate of postoperative plasma ctDNA methylation-MRD detection results for 2-year tumor recurrence rate after colorectal cancer radical resection was calculated.
- MRD negative group: ColonAiQ polygene methylation test was performed on peripheral blood plasma samples from the enrolled patients 4 weeks after surgery. If the gene methylation level detected in the samples did not exceed the threshold, the patients were enrolled in the MRD negative group. The 2-year total tumor recurrence rate of patients in the negative MRD group was calculated, and the negative prediction rate of postoperative plasma ctDNA methylation-MRD test results for 2-year tumor recurrence rate after radical resection of colorectal cancer was calculated.

SUMMARY:
This study dynamically monitored the prognosis of stage I-IV colorectal cancer patients who could receive radical surgical resection by detecting the levels of polygene methylation in plasma samples from patients with colorectal cancer. In patients with colorectal cancer feasible radical surgery, plasma ctDNA methylation detection was performed before and after surgical treatment and during regular follow-up to explore the predictive effect of plasma ctDNA methylation status at different time points on postoperative recurrence. To explore whether postoperative dynamic monitoring of plasma ctDNA methylation can be used for adjuvant chemotherapy efficacy evaluation and whether it can indicate tumor recurrence and metastasis earlier than imaging examination.

DETAILED DESCRIPTION:
1. Patients initially diagnosed with primary colorectal cancer were enrolled for screening, and plasma samples 1-2 days before radical bowel resection were collected for polygene methylation detection.
2. The postoperative follow-up was 2 years, and the reexamination included CT/MRI imaging assessment, blood CEA, and dynamic monitoring of plasma ctDNA methylation level. Blood samples were collected for 9 times.
3. Results analysis: To explore the application value of ctDNA methylation-MRD detection in the prediction of postoperative tumor recurrence risk after radical resection of colorectal cancer; The correlation between preoperative ctDNA methylation level and prognosis of early colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed patients with primary colorectal cancer confirmed by histopathology (no restriction on histological type);
2. Patients diagnosed as stage I-III and feasible for radical bowel surgery;
3. Patients diagnosed by stage IV (only colorectal cancer patients with liver metastasis at the time of diagnosis) and feasible radical bowel resection or complete resection of liver metastasis;
4. No gender limitation, age ≥18;
5. ECOG score ≤1;
6. Life expectancy ≥5 years;
7. Those who fully understand the study and voluntarily sign the informed consent.

Exclusion Criteria:

1. Blood transfusion was performed during surgery or 2 weeks before surgery;
2. complicated with primary malignant tumors of other organs;
3. With colonic obstruction, intestinal perforation and other symptoms requiring emergency treatment;
4. Colorectal cancer was diagnosed with extrahepatic metastasis;
5. Neoadjuvant therapy (such as radiotherapy and chemotherapy) before radical bowel resection;
6. Radical bowel resection was performed after endoscopic surgery;
7. Concomitant symptoms and/or family history collection suggest hereditary colorectal cancer;
8. serious mental illness or drug abuse;
9. patients with serious heart, lung and vascular diseases who cannot tolerate surgery;
10. pregnant or lactating women;
11. Participate in other interventional clinical investigators within 3 months
12. Poor compliance, unable to complete the study according to the judgment of the researcher.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 800 patients with initial clinical diagnosis of primary colorectal cancer
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2022-06-20 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
To establish a clinical cohort for colorectal cancer | assessed up to 36 months
  It is expected that 800 patients with primary colorectal cancer diagnosed clinically will be enrolled for screening. Plasma samples 1-2 days before radical bowel resection will be collected for ColonAiQ polygene methylation test. Follow-up will be conducted 2 years after surgical resection, including CT/MRI imaging evaluation and blood CEA, etc. And dynamic monitoring of plasma ctDNA methylation level. Blood samples were collected for 9 times.
To investigate the prediction and monitoring effect of plasma ctDNA methylation on postoperative recurrence of primary colorectal cancer patients after radical surgery | assessed up to 36 months
  To investigate the role of peripheral plasma ctDNA methylation level at different time points in the monitoring of disease recurrence after radical bowel resection for primary colorectal cancer, the multi-gene methylation detection of peripheral plasma ctDNA was conducted before, after and during the postoperative follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Rui Liu, Doctor, Principal Investigator — Singlera Genomics Inc.
Locations (7):
- China (7):
  - Cancer hospital Chinese academy of medical sciences, Beijing, Beijing Municipality
  - West China Hospital, Chengdu
  - Sun Yat-sen University Cancer Center, Guangzhou
  - The Second Affiliated Hospital of Harbin Medical University, Haerbin
  - The First Affiliated Hospital of Naval Medical University/ Changhai Hospital, Shanghai
  - Chinese Academy of Medical Sciences, Shenzhen Center, Shenzhen
  - Shanxi Cancer hospital (Shanxi Cancer institute), Taiyuan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Young PE, Womeldorph CM, Johnson EK, Maykel JA, Brucher B, Stojadinovic A, Avital I, Nissan A, Steele SR. Early detection of colorectal cancer recurrence in patients undergoing surgery with curative intent: current status and challenges. J Cancer. 2014 Mar 15;5(4):262-71. doi: 10.7150/jca.7988. eCollection 2014. PMID 24790654
- [Background] Pantel K, Alix-Panabieres C. Tumour microenvironment: informing on minimal residual disease in solid tumours. Nat Rev Clin Oncol. 2017 Jun;14(6):325-326. doi: 10.1038/nrclinonc.2017.53. Epub 2017 Apr 11. No abstract available. PMID 28397823